CLINICAL TRIAL: NCT03371862
Title: Pilot Study of the GLP-1 Agonist, Liraglutide, on Decreasing Parenteral Support Requirements in Short Bowel Patients.
Brief Title: Liraglutide on Decreasing Parenteral Support in Short Bowel Patients (SLIPS)
Acronym: SLIPS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants recruited. Not able to recruit due to COVID 19.
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17IC3834
Record Dates: First submitted 2017-10-25; First posted 2017-12-13 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Short Bowel Syndrome
Keywords: Liraglutide; Victoza
MeSH Terms: conditions — Short Bowel Syndrome | interventions — Liraglutide

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Test group (Experimental)
  Interventions: Drug: Liraglutide Pen Injector [Victoza]

INTERVENTIONS:
Drug: Liraglutide Pen Injector [Victoza] — Pilot study of liraglutide in patients with short bowel.

SUMMARY:
Pilot study looking at the effect on Liraglutide in the reduction of parenteral support in patients with short bowel.

ELIGIBILITY:
Inclusion Criteria:

1. Short bowel (≤200cm) as a result of major intestinal resection (e.g. due to injury, volvulus, vascular disease, Crohn's disease).
2. Jejunostomy patients only
3. 12 continuous months of parenteral support (PS) dependency prior to enrolment.
4. PS required at least 3 times per week to meet their caloric, fluid or electrolyte needs due to on-going malabsorption.
5. Stable PS for at least 4 consecutive weeks immediately prior to first dose of liraglutide. Stability is described as:

   1. Actual PS usage should match prescribed PS;
   2. Baseline 48-hour urine output is 1-2 L/24 hours.
6. Body mass index ≥ 19.5 kg/m2.
7. Adequate hepatic and renal function:

   1. Total bilirubin within the normal range;
   2. Alanine aminotransferase (ALT) ≤ 2.5x upper limit of normal;
   3. Serum creatinine ≤1.5x upper limit of normal.
8. Stable dosage for > 4 weeks, prior to baseline evaluations, of anti-motility and anti-diarrhoeal agents, H2 antagonists, proton pump inhibitors, bile sequestering agents and oral rehydration solutions.
9. Female subjects must be on acceptable method of contraception for a minimum of 4 weeks prior to the start of the trial; Acceptable methods of contraception would be a barrier form of contraception, oral contraceptive pill, contraceptive injection or implant or intrauterine implanted device.

Exclusion Criteria:

* Patients < 18 years of age
* Pregnancy (Female subjects who are not surgically sterile or post menopausal (defined as aged 55 years or older and/or at least 2 years have elapsed since the last menses) or who are not using medically acceptable methods of birth control during and for 30 days after the treatment period. Acceptable methods of contraception would be a barrier form of contraception, oral contraceptive pill, contraceptive injection or implant or intrauterine implanted device.
* Active malignancy
* Previous malignancy within the past 5 years
* History of multiple endocrine neoplasia type 2 (MEN 2)
* Personal history or family history of medullary thyroid cancer
* Raised serum calcitonin (a biomarker for medullary thyroid cancer) at beginning of trial period
* History of cardiac failure
* Concurrent use of diuretics
* Previous history of pancreatitis
* Recent use of other incretin based therapy in the previous 3 months
* Concurrent use of octreotide
* Type 1 or Type 2 diabetes
* Alcohol or drug abuse in last year
* > 4 hospitalisations related to short bowel or its treatment over the previous year
* Any hospitalisation 30 days prior to screening
* Introduction or dose adjustment of immunosuppressant for inflammatory bowel disease within 6 months, or treatment with biologics within the past 6 months (systemic corticosteroids, methotrexate, cyclosporine, tacrolimus, sirolimus, MMF, infliximab, adalimumab, vedolizumab)
* BMI < 19 kg/m2 or > 27kg/m2 (An upper cut-off BMI of > 27kg/m2 has been chosen, as in these patients, there is often a desire to reduce BMI which will conflict with the study design by adding another variable)
* Scleroderma/radiation enteritis/coeliacs disease/refractory or tropical sprue
* Liver and renal function outside the inclusion range

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in parenteral support | 20 weeks post start of drug
  Improvement of parenteral support on 20 weeks of Liraglutide

SECONDARY OUTCOMES:
Improvement in quality of life | 20 weeks post start of drug
  Improvement in Euroqol EQ5-D score. Level 1: indicating no problem, Level 5: indicating extreme problems.
Duration of response | 20 weeks
  Duration of response i.e. proportion of subjects who maintain reduction in weekly PN volume from baseline at week 20.
Days/Nights not requiring PS | 20 weeks
  Days/Nights not requiring PS
Change in plasma citrulline, GLP-1, IGF-1 and PYY concentrations | 20 weeks
  Change in plasma citrulline, GLP-1, IGF-1 and PYY concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Siddhartha Oke, Principal Investigator — Imperial College London
Locations (1):
- St Mark's Hospital, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided